CLINICAL TRIAL: NCT04540042
Title: A Two Part, Randomised, Double-blind, Placebo-controlled, Phase 2 Parallel Group Study to Evaluate the Safety and Efficacy of Intravenously-Administered SelK2 on Airway Responses Following Allergen Challenge in Subjects With Asthma (Part 1) and to Evaluate the Safety and Efficacy of Intravenously-Administered SelK2 in Subjects With Chronic Obstructive Pulmonary Disease (Part 2)
Brief Title: Study to Assess the Safety and Efficacy of SelK2 on Airway Responses Following Allergen Challenge in Subjects With Asthma (Part 1) and in Subjects With Chronic Obstructive Pulmonary Disease (Part 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tetherex Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SELK2-00006; 2020-001027-13 (EudraCT Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: asthma; chronic obstructive pulmonary disease; COPD; adhesion molecule; P-selectin glycoprotein ligand 1; P-selectin
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Part 1 of the study will enroll patients in two arms in a 1:1 ratio to receive either SelK2 or placebo. Part 2 of the study will enroll patients in two arms in a 2:1 ratio to receive either SelK2 or placebo, respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SelK2 (Part 1) (Experimental): I.V., multiple-dose (Day 1 and Day 22)
  Interventions: Drug: SelK2 (Part 1)
- Placebo (Part 1) (Placebo Comparator): I.V., multiple-dose (Day 1 and Day 22)
  Interventions: Drug: Placebo (Part 1)
- SelK2 (Part 2) (Experimental): I.V., single-dose (Day 1)
  Interventions: Drug: SelK2 (Part 2)
- Placebo (Part 2) (Placebo Comparator): I.V., single-dose (Day 1)
  Interventions: Drug: Placebo (Part 2)

INTERVENTIONS:
Drug: SelK2 (Part 1) — I.V., multiple-dose (Day 1 and Day 22)
  Arms: SelK2 (Part 1)
Drug: Placebo (Part 1) — I.V., multiple-dose (Day 1 and Day 22)
  Arms: Placebo (Part 1)
Drug: SelK2 (Part 2) — I.V., single-dose (Day 1)
  Arms: SelK2 (Part 2)
Drug: Placebo (Part 2) — I.V., single-dose (Day 1)
  Arms: Placebo (Part 2)

SUMMARY:
This study has two parts. The main purpose of Part 1 of this study will be to examine how safe and effective two doses of SelK2 is on participants with mild asthma. Lung function and inflammatory cell numbers will be measured in response to the administration of an allergen (a compound to which the participant is allergic) into the lungs in the presence or absence of SelK2. Part 2 of this study will examine how safe and effective one dose of SelK2 is on participants with chronic obstructive pulmonary disease (COPD). Lung function and inflammatory cell numbers will be measured in COPD patients in the presence or absence of SelK2. SelK2 may block the movement of key inflammatory cells into the lungs and consequently improve lung function in these two patient populations.

ELIGIBILITY:
Part 1:

Key Inclusion Criteria

* Males or females, 18-65 years of age (inclusive)
* Body Mass Index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2
* Documented physician-diagnosed asthma for ≥ 4 months prior to screening
* Pre-bronchodilator FEV1 ≥ 70% predicted at screening
* Documented allergy to at least one common allergen as confirmed by the skin prick test
* Dual responder to inhaled bronchial allergen challenges as manifested by positive allergen-induced early (EAR) and late airway bronchoconstriction (LAR) at screening

Key Exclusion Criteria

* Lung disease other than stable, mild asthma; e.g., worsening of asthma that requires a change in asthma therapy in the past 4 weeks or is deemed clinically significant by the investigator.
* A diagnosed current or recent (within previous 8 weeks of screening, or prior to randomisation) bacterial, protozoal, viral or parasitic infection; is suspected of or is at high risk of having a parasitic infection, or has a history of more than one episode of herpes zoster infection.
* Has a history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest and/or hypoxic seizures.
* Has been hospitalised or has attended the emergency room for asthma in the 12 months prior to screening, or prior to randomisation.
* A history of tuberculosis (latent or active) or systemic fungal diseases.

Part 2:

Key Inclusion Criteria

* Male or female, 40 to 75 years of age, inclusive, at the time of informed consent.
* Confirmed diagnosis by a physician of COPD with symptoms compatible with COPD for at least 1 year prior to screening.
* BMI ≥ 18.0 and ≤ 35.0 kg/m2 at screening.
* Able to tolerate sputum induction and produce an adequate sputum sample with a neutrophil differential count > 55% at screening.
* Post-bronchodilator FEV1 ≥ 30% and ≤ 80% of the predicted normal, and post-bronchodilator FEV1/FVC < 0.7 at the time of Screening.
* Current or former tobacco smoker who has a smoking history of at least 10 pack years (Ten pack- years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years).
* Has a negative result in the blood test for tuberculosis (TB) at screening.

Key Exclusion Criteria

* COPD exacerbation requiring oral steroids and/or antibiotics, within the 8 weeks prior to screening or prior to randomisation.
* A positive sputum culture at Screening indicating ongoing infection.
* Other respiratory disorders: Subjects with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, known alpha-1 antitrypsin deficiency or other active pulmonary diseases other than COPD.
* A history of life-threatening COPD including intensive care unit admission and/or requiring intubation within the last 5 years.
* A history of > 1 hospitalisation for COPD in the previous 1 year prior to screening.
* Previous lung resection, lung reduction surgery or lung transplantation.
* Requires supplemental oxygen, even on an occasional basis.
* Any infection requiring hospitalisation or intravenous antibiotics within 6 months prior to Screening or prior to randomisation.
* A diagnosed current or recent (within previous 8 weeks of screening, or prior to randomisation) bacterial, protozoal, viral or parasitic infection; is suspected of or is at high risk of having a parasitic infection, or has a history of more than one episode of herpes zoster infection.
* Active participation in a pulmonary rehabilitation program.
* A history of tuberculosis (latent or active) or systemic fungal diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum percentage fall in FEV1 from pre-challenge between 3 and 8 hours (LAR) after administration of allergen inhalation challenge (Part 1). | Pre-challenge to between 3 and 8 hours after administration of allergen inhalation challenge
Change from baseline in percentage of neutrophils in sputum (Part 2). | Change from baseline to Day 22

SECONDARY OUTCOMES:
AUC for the percent fall in FEV1 from pre-challenge between 3 and 8 hours (LAR) after the administration of allergen inhalation challenge (Part 1). | Pre-challenge to between 3 and 8 hours after administration of allergen inhalation challenge
Change from baseline and change during challenge in percentage of eosinophils in sputum (Part 1) | Change from baseline to 8 and 24 hours post allergen challenge
Maximum percentage fall in FEV1 and AUC for the percent fall in FEV1 from pre-challenge between 0 and 2 hours after the administration of allergen inhalation challenge (EAR) (Part 1). | Pre-challenge to between 0 and 2 hours after the administration of allergen inhalation challenge
Maximum percentage fall in FEV1 and AUC for the percent fall in FEV1 between 0 and 8 hours (entire asthmatic response) after the administration of allergen inhalation challenge (Part 1) | Pre-challenge to between 0 and 8 hours after the administration of allergen inhalation challenge
Change from baseline in pre-challenge FEV1 (Part 1). | Change from baseline to Day 29
Change from baseline in percentage of neutrophils (Part 2). | Change from baseline to Days 4, 8, 15, and 29
Change from baseline in absolute and percentage cell counts for immune cells in induced sputum samples and blood (Part 2). | Change from baseline to Days 4, 8, 15, 22, and 29
Change from baseline in FEV1 and post-bronchodilator FEV1 (Part 2). | Change from baseline to Days 4, 8, 15, 22, and 29
Change from baseline in pre- and post-bronchodilator impulse oscillometry (IOS) (Part 2). | Change from baseline to Days 4, 8, 15, 22, and 29
Change from baseline in pre- and post-bronchodilator whole body plethysmography (Part 2). | Change from baseline to Days 4, 8, 15, 22, and 29
Change from baseline in COPD Assessment Test (CAT) scores (Part 2). | Change from baseline to Days 4, 8, 15, 22, and 29
  Scores range from 0-40 with 40 being associated with the worst outcome.
Change from baseline in Breathlessness Cough and Sputum Scale (BCSS) scores (Part 2). | Change from baseline to Days 4, 8, 15, 22, and 29
  Scores range from 0-12 with 12 being associated with the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Stocker, Ph.D., Study Director — Tetherex Pharmaceuticals Corporation
Locations (2):
- United Kingdom (2):
  - Queen Anne Street Medical Centre, London
  - Medicines Evaluation Unit Ltd., Manchester